CLINICAL TRIAL: NCT02869841
Title: Efficacy of Rectal Sheath Analgesia After Midline Laparotomy
Acronym: Rektus-puu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-14
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2020-08

CONDITIONS: Surgery; Pain Postoperative
Keywords: laparotomy; pain; rectus sheath block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Continuous rectus sheath analgesia (Active Comparator): Local anesthetic continuous infusion with infusion pumps
  Interventions: Drug: Levobupivacaine continuous infusion
- Bolus rectus sheath analgesia (Active Comparator): Bolus administration of local anesthetic
  Interventions: Drug: levobupivacaine bolus dosing
- Single dose rectus sheath analgesia (Active Comparator): single dose administration of local anesthetic
  Interventions: Drug: single bolus of levobupivacaine
- Placebo (Placebo Comparator): no rectus sheath analgesia
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levobupivacaine continuous infusion — Levobupivacaine continuous infusion to rectus sheath catheters
  Other Names: continuous infusion group
  Arms: Continuous rectus sheath analgesia
Drug: levobupivacaine bolus dosing — Levobupivacaine bolus dosing to rectus sheath catheters
  Other Names: bolus group
  Arms: Bolus rectus sheath analgesia
Drug: single bolus of levobupivacaine — Levobupivacaine single dose to rectus sheath catheters
  Other Names: single dose group
  Arms: Single dose rectus sheath analgesia
Other: Placebo — No rectus sheath analgesia
  Other Names: no rectus sheath catheters
  Arms: Placebo

SUMMARY:
Midline laparotomy is commonly used in emergency and elective cancer surgery and patients need effective and safe pain treatment after this type of surgery. Nowadays modern anticoagulant therapy may prevent use of central regional blocks in pain management. Therefore in the present study the efficacy and safety of rectus sheath analgesia is studied using different administration techniques. The primary aim is the efficacy of the rectus sheath analgesia measured with pain ratings and the amount rescue opioid used.

Secondary aims were concentrations of local anesthetic, rescue opioid and satisfaction to analgesia method used.

ELIGIBILITY:
Inclusion Criteria: • Body mass index over BMI <35 kg / m2

* not pregnancy/adequate contraception
* no contraindications to the local anaesthetic No contraindications to opioid patient controlled analgesia
* Informed consent obtained

Exclusion Criteria:

* • BMI >35 kg / m2

  * Pregnant or breast feeding
  * Contraindication to local anaesthetics
  * Contraindication to opioids
  * Not able to use patient controlled analgesia pump
  * Relaparotomy
  * No informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2018-07 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Amount of rescue analgesic used for pain relief | Time 0 h up to 48 h postoperatively
  From onset of rectus sheath analgesia

SECONDARY OUTCOMES:
Maximum levobupivacaine plasma concentration | Time 0 h to 48 h postoperatively
  Maximum levobupivacaine plasma concentration
maximum rescue analgesic concentration | time 0 h to 48 h postoperatively
  maximum rescue analgesic concentration

CONTACTS AND LOCATIONS:
Overall Officials: Matti Eskelinen, Professor, Study Chair — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No